CLINICAL TRIAL: NCT02187861
Title: A Phase II, Open-Label Study Evaluating the Safety and Efficacy of GDC-0199 (ABT-199) Plus Bendamustine Plus Rituximab (BR) in Comparison With BR Alone or GDC-0199 Plus Rituximab (R) in Patients With Relapsed and Refractory Follicular Non-Hodgkin's Lymphoma
Brief Title: A Study Evaluating the Safety and Efficacy of Venetoclax (GDC-0199) Plus Bendamustine + Rituximab (BR) in Comparison With BR or Venetoclax Plus Rituximab in Participants With Relapsed and Refractory Follicular Non-Hodgkin's Lymphoma (fNHL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO29337; 2014-000576-26 (EudraCT Number)
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — venetoclax; Bendamustine Hydrochloride; Rituximab

ARMS (4):
- Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) (Experimental): Participants will receive venetoclax no more than 600 milligrams (mg) orally once daily continuously along with rituximab 375 milligrams per square meter (mg/m^2) intravenous (IV) infusion on Day 1 of 28-day cycle and bendamustine 90 mg/m^2 IV infusion on Days 1 and 2 of the 28-day cycle. Safety run-in will continue until first 9 participants complete the safety observation window of 28 days. Participants will continue receiving the same treatment as decided for Arm B.
  Interventions: Drug: Venetoclax; Drug: Bendamustine; Drug: Rituximab
- Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) (Experimental): Participants will receive venetoclax 800 mg orally once daily for 1 year along with rituximab 375 mg/m^2 IV infusion on Days 1, 8, 15, 22 of Cycle 1 and Day 1 of Cycles 4, 6, 8, 10, and 12. Each cycle will be of 28 days.
  Interventions: Drug: Venetoclax; Drug: Rituximab
- Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) (Experimental): Participants will receive venetoclax at doses decided from safety run-in orally once daily continuously for 1 year along with rituximab 375 mg/m^2 IV infusion on Day 1 of each 28-day cycle and bendamustine 90 mg/m^2 IV infusion on Days 1 and 2 of each 28-day cycle, for 6 cycles.
  Interventions: Drug: Venetoclax; Drug: Bendamustine; Drug: Rituximab
- Chemotherapy-Containing Cohort: Arm C (BR) (Active Comparator): Participants will receive rituximab 375 mg/m^2 IV infusion on Day 1 of each 28-day cycle and bendamustine 90 mg/m^2 IV infusion on Days 1 and 2 of each 28-day cycle, for 6 cycles.
  Interventions: Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Venetoclax — Venetoclax will be administered as per the schedule specified under arm description.
  Other Names: GDC-0199; ABT-199
  Arms: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR); Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR); Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab)
Drug: Bendamustine — Bendamustine will be administered as per the schedule specified under arm description.
  Other Names: Levact
  Arms: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR); Chemotherapy-Containing Cohort: Arm C (BR); Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR)
Drug: Rituximab — Rituximab will be administered as per the schedule specified under arm description.
  Other Names: MabThera; Rituxan

SUMMARY:
This open-label, international, multicenter study will investigate the safety and efficacy of venetoclax (GDC-0199) in combination with bendamustine plus rituximab (venetoclax + BR) compared with BR alone in participants with relapsed and refractory fNHL, comparing two chemotherapy-containing regimens (Chemotherapy-Containing Cohort). In addition, an exploratory analysis of the safety and efficacy of venetoclax in combination with rituximab (venetoclax + rituximab), a chemotherapy-free regimen, will be performed (Chemotherapy-Free Cohort). Assignment to the Chemotherapy-Containing or Chemotherapy-Free Cohort will be decided at the discretion of the Investigator, unless one of the cohorts is not open to enrollment; in which case, participants may be enrolled only to the open cohort. The first 6 participants enrolled in the Chemotherapy-Containing Cohort (or more if required) will comprise the Safety Run-In group for Treatment Arm B, dosing venetoclax at 600 milligrams (mg) in combination with BR. Once a dose has been chosen from the Safety Run-In Period, randomization to the two treatment arms of the Chemotherapy-Containing Cohort (Arms B and C) will begin.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed follicular lymphoma (FL) of Grade 1, 2, or 3a
* Participants must have received at least one prior therapy for FL
* For participants potentially receiving chemotherapy: if the participant has received prior bendamustine, response duration must have been greater than (>) 1 year
* At least one bi-dimensionally measurable lesion on imaging scan defined as >1.5 centimeters (cm) in its longest dimension
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Adequate hematologic function
* For female participants of childbearing potential and male participants with female partners of childbearing potential, agreement to use one highly effective form of non-hormonal contraception or two effective forms of non-hormonal contraception throughout the course of study treatment and for at least 30 days after the last dose of venetoclax and 12 months after the last dose of rituximab, whichever is longer
* Confirmed availability of archival or freshly biopsied tumor tissue meeting protocol-defined specifications prior to study enrollment

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
* Contraindication to potential treatment agents
* Ongoing corticosteroid use >30 milligrams per day (mg/day) of prednisone or equivalent. Participants receiving corticosteroid treatment with less than equal to (</=) 30 mg/day of prednisone or equivalent must be documented to be on a stable dose of at least 4 weeks duration prior to randomization (Cycle 1 Day 1)
* Primary central nervous system (CNS) lymphoma
* Vaccination with live vaccines within 28 days prior to treatment
* Chemotherapy or other investigational therapy within five half-lives of a biologic agent with a minimum of 28 days prior to the start of Cycle 1
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results or that could increase risk to the participant
* Significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, congestive heart failure, myocardial infarction within the previous 6 months, unstable arrhythmias, or unstable angina) or significant pulmonary disease (including obstructive pulmonary disease and history of bronchospasm)
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection requiring treatment with intravenous antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1 Day 1
* Requires the use of warfarin
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Presence of positive test results for hepatitis B surface antigen or hepatitis C virus (HCV) antibody
* Participants who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation
* Participants with occult or prior hepatitis B virus (HBV) infection may be included if HBV deoxyribonucleic acid (DNA) is undetectable at screening. These participants must be willing to undergo monthly HBV DNA test until at least 12 months after the last treatment cycle
* Known infection with human immunodeficiency virus (HIV) or human T-cell leukemia virus 1 (HTLV-1)
* Pregnant or lactating
* Recent major surgery (within 6 weeks before the start of Cycle 1 Day 1), other than for diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2018-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (71):
- United States (17):
  - Southern Cancer Center, PC, Mobile, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - UCLA School of Medicine; Hematology/Oncology, Los Angeles, California
  - Nothwest Georgia Oncology Centers P.C, Austell, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago College of Medicine, Chicago, Illinois
  - Primary Healthcare Associates SC - Harvey, Harvey, Illinois
  - University of Kansas; Medical Center & Medical pavilion, Westwood, Kansas
  - Sidney Kimmel Comp Cancer Ctr, Baltimore, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey
  - James P. Wilmot Cancer Center, Rochester, New York
  - University of Pennsylvania; School of Medicine, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - VCU Massey Cancer Center, Richmond, Virginia
  - West Virginia Uni Med. Center - Robert Byrd Health Science, Morgantown, West Virginia
- Australia (10):
  - Royal Prince Alfred Hospital; Medical Oncology, Camperdown, New South Wales
  - St George Hospital, Kogarah, New South Wales, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital; Haematology, Sydney, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Townsville General Hospital, Douglas, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Queen Elizabeth Hospital; Haematology, Woodville South, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre, Clayton, Victoria
- Belgium (3):
  - ZNA Stuivenberg, Antwerp
  - AZ Sint Jan, Bruges
  - Cliniques Universitaires St-Luc, Brussels
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Kelowna, British Columbia
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
  - Hopital Maisonneuve- Rosemont; Oncology, Montreal, Quebec
  - Chum Hopital Notre Dame; Centre D'Oncologie, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Saskatoon Cancer Centre; Uni of Saskatoon Campus, Saskatoon, Saskatchewan
- France (7):
  - Institut de Cancerologie de l'Ouest, Angers
  - CHU Clermont Ferrand - Hôpital d'Estaing, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - CHU de Dijon - Hopital le Bocage, Dijon
  - Centre Jean Bernard, Le Mans
  - CHU Montpellier, Montpellier
  - Centre Hospitalier Lyon Sud; Hematolgie, Pierre-Bénite
- Germany (10):
  - Klinikum Chemnitz gGmbH; Klinik f. Innere Medizin III, Chemnitz
  - Universitätsklinikum Köln; Klinik I für Innere Medizin, Cologne
  - Städtisches Klinikum Dessau, Dessau
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf; Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Universitätsklinik Essen; Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Essen
  - Universitätsklinikum Jena; Klinik für Innere Medizin II, Jena
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck, Med. Klinik I, Hämatologie/Onkologie, Lübeck
  - Uni. der Johannes Gutenberg-Universitaet Mainz; III. Medizinische Klinik und Poliklinik, Mainz
  - Universitätsklinikum Ulm; Apotheke, Ulm
  - Universitätsklinikum Würzburg; Medizinische Klinik und Poliklinik II; Hämatologie / Onkologie, Würzburg
- Italy (9):
  - A.O. Universitaria Policlinico S.Orsola-Malpighi Di Bologna, Bologna, Emilia-Romagna
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Ospedale di Ravenna, Ravenna, Emilia-Romagna
  - Ospedale Infermi di Rimini, Rimini, Emilia-Romagna
  - Asst Papa Giovanni XXIII, Bergamo, Lombardy
  - Ospedale Niguarda Milano, Milan, Lombardy
  - Irccs Policlinico San Matteo; Divisione Di Ematologia, Pavia, Lombardy
  - Azienda Ospedale San Giovanni, Turin, Piedmont
  - Az. Osp. Di Careggi; Divisione Di Ematologia, Florence, Tuscany
- United Kingdom (8):
  - Blackpool Victoria Hospital, Blackpool
  - St James University Hospital, Leeds
  - Leicester Royal Infirmary; Dept. of Medical Oncology, Leicester
  - University College London, Department of Haematology, London
  - Royal Marsden Nhs Trust; Consultant Cancer Physician, London
  - Christie Hospital; Breast Cancer Research Office, Manchester
  - Churchill Hospital; Oxford Cancer and Haematology Centre, Oxford
  - Royal Marsden NHS Foundation Trust, Sutton

REFERENCES:
- [Derived] Zinzani PL, Flinn IW, Yuen SLS, Topp MS, Rusconi C, Fleury I, Le Du K, Arthur C, Pro B, Gritti G, Crump M, Petrich A, Samineni D, Sinha A, Punnoose EA, Szafer-Glusman E, Spielewoy N, Mobasher M, Humphrey K, Kornacker M, Hiddemann W. Venetoclax-rituximab with or without bendamustine vs bendamustine-rituximab in relapsed/refractory follicular lymphoma. Blood. 2020 Dec 3;136(23):2628-2637. doi: 10.1182/blood.2020005588. PMID 32785666

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR): Participants received venetoclax no more than 600 milligrams (mg) orally once daily continuously along with rituximab 375 milligrams per square meter (mg/m^2) intravenous (IV) infusion on Day 1 of 28-day cycle and bendamustine 90 mg/m^2 IV infusion on Days 1 and 2 of the 28-day cycle. Safety run-in continued until first 9 participants completed the safety observation window of 28 days. After first 28 days of safety observation (Cycle 1), participants continued to receive venetoclax 600 mg orally once daily up to 1 year along with rituximab 375 mg/m^2 IV infusion on Day 1 of each 28-day cycle and bendamustine 90 mg/m^2 IV infusion on Days 1 and 2 of each 28-day cycle, for 6 cycles.
- Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab): Participants received venetoclax 800 mg orally once daily for 1 year along with rituximab 375 mg/m^2 IV infusion on Days 1, 8, 15, 22 of Cycle 1 and Day 1 of Cycles 4, 6, 8, 10, and 12. Each cycle was of 28 days.
- Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR): Participants received venetoclax 800 mg orally once daily continuously for 1 year along with rituximab 375 mg/m^2 IV infusion on Day 1 of each 28-day cycle and bendamustine 90 mg/m^2 IV infusion on Days 1 and 2 of each 28-day cycle, for 6 cycles.
- Chemotherapy-Containing Cohort: Arm C (BR): Participants received rituximab 375 mg/m^2 IV infusion on Day 1 of each 28-day cycle and bendamustine 90 mg/m^2 IV infusion on Days 1 and 2 of each 28-day cycle, for 6 cycles.
Period: Overall Study
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Started | 9 | 52 | 51 | 51
Treated | 9 | 52 | 49 | 50
Completed | 3 | 4 | 19 | 19
Not Completed | 6 | 48 | 32 | 32
Not completed — Adverse Event | 2 | 1 | 2 | 1
Not completed — Death | 0 | 3 | 1 | 2
Not completed — Physician Decision | 0 | 1 | 0 | 3
Not completed — Progressive Disease | 4 | 42 | 19 | 22
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 3
Not completed — Other | 0 | 1 | 7 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR) | Total
Number analyzed (Participants) | 9 | 52 | 51 | 51 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (12.7) | 61.9 (12.0) | 64.9 (9.8) | 61.0 (11.6) | 62.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 25 | 16 | 21 | 67
  Male | 4 | 27 | 35 | 30 | 96

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Metabolic Response (CMR) According to Independent Review Committee (IRC) as Per Lugano Classification, Using Positron Emission Tomography (PET) Scan at Primary Response Assessment (PRA)
Description: CMR: a score 1 (no uptake above background), 2 (uptake less than or equal to [<=] mediastinum), or 3 (uptake less than [<] mediastinum but <=liver) with or without a residual mass on PET 5-point scale (5-PS), for lymph nodes and extralymphatic sites with no new lesions and no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow. Assessment was performed by an IRC according to Lugano classification using PET scan. 95% confidence interval (CI) for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 6-8 weeks after Cycle 6 Day 1 (PRA) (Cycle length = 28 days)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
percentage of participants | 55.6 [21.20 to 86.30] | 11.5 [4.35 to 23.44] | 74.5 [60.37 to 85.67] | 70.6 [56.17 to 82.51]
Statistical Analysis 1: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); Test type: Superiority or Other; Difference in response rates = 3.92, 95% CI 2-sided [-13.38 to 21.23]

2. Secondary Outcome: Percentage of Participants With CMR According to Investigator as Per Lugano Classification, Using PET Scan at PRA
Description: CMR: a score 1 (no uptake above background), 2 (uptake <=mediastinum), or 3 (<mediastinum but <=liver) with or without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites with no new lesions and no evidence of FDG-avid disease in bone marrow. Assessment was performed by Investigator according to Lugano classification using PET scan. 95% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 4-10 weeks after Cycle 6 Day 1 (Cycle length = 28 days)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
percentage of participants | 55.6 [21.20 to 86.30] | 15.4 [6.88 to 28.08] | 70.6 [56.17 to 82.51] | 68.6 [54.11 to 80.89]
Statistical Analysis 1: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); Test type: Superiority or Other; Difference in response rates = 1.96, 95% CI 2-sided [-15.89 to 19.81]

3. Secondary Outcome: Percentage of Participants With CMR According to IRC as Per Lugano Classification, Using PET Scan at Year 1
Description: CMR: a score 1 (no uptake above background), 2 (uptake <=mediastinum), or 3 (uptake <mediastinum but <=liver) with or without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites with no new lesions and no evidence of FDG-avid disease in bone marrow. Assessment was performed by an IRC according to Lugano classification using PET scan. 95% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 48-56 weeks after Cycle 1 Day 1 (Cycle length = 28 days)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
percentage of participants | 55.6 [21.20 to 86.30] | 21.2 [11.06 to 34.70] | 41.2 [27.58 to 55.83] | 39.2 [25.84 to 53.89]
Statistical Analysis 1: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); Test type: Superiority or Other; Difference in response rates = 1.96, 95% CI 2-sided [-17.07 to 20.99]

4. Secondary Outcome: Percentage of Participants With CMR According to Investigator as Per Lugano Classification, Using PET Scan at Year 1
Description: as for outcome 2
Time Frame: 48-56 weeks after Cycle 1 Day 1 (Cycle length = 28 days)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
percentage of participants | 55.6 [21.20 to 86.30] | 17.3 [8.23 to 30.33] | 39.2 [25.84 to 53.89] | 47.1 [32.93 to 61.54]
Statistical Analysis 1: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); Test type: Superiority or Other; Difference in response rates = -7.84, 95% CI 2-sided [-27.01 to 11.32]

5. Secondary Outcome: Percentage of Participants With Complete Response (CR) According to IRC as Per Lugano Classification, Using Computed Tomography (CT) Scan
Description: CR: defined as reduction of longest transverse diameter of lesion (LDi) of target nodes/nodal masses to <=1.5 centimeters (cm), and no extralymphatic sites of disease; absence of non-measured lesions and new lesions; reduction of enlarged organs to normal; and normal/immunohistochemistry (IHC)-negative bone marrow morphology. Assessment was performed by an IRC according to Lugano classification using CT scan. 95% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 6-8 weeks after Cycle 6 Day 1 and 48-56 weeks after Cycle 1 Day 1 (Cycle length = 28 days)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
percentage of participants
  6-8 weeks after Cycle 6 Day 1 | 44.4 [13.70 to 78.80] | 5.7 [1.18 to 15.66] | 39.2 [25.84 to 53.89] | 25.5 [14.33 to 39.63]
  Year 1 | 55.6 [21.20 to 86.30] | 13.2 [5.48 to 25.34] | 27.5 [15.89 to 41.74] | 23.5 [12.79 to 37.49]
Statistical Analysis 1: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); At 6-8 weeks after Cycle 6 Day 1; Test type: Superiority or Other; Difference in response rates = 13.73, 95% CI 2-sided [-4.24 to 31.69]
Statistical Analysis 2: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); At Year 1; Test type: Superiority or Other; Difference in response rates = 3.92, 95% CI 2-sided [-12.98 to 20.82]

6. Secondary Outcome: Percentage of Participants With CR According to Investigator as Per Lugano Classification, Using CT Scan
Description: CR: defined as reduction of LDi of target nodes/nodal masses to <=1.5 cm, and no extralymphatic sites of disease; absence of non-measured lesions and new lesions; reduction of enlarged organs to normal; and normal/IHC-negative bone marrow morphology. Assessment was performed by Investigator according to Lugano classification using CT scan. 95% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 4-10 weeks after Cycle 6 Day 1 and 48-56 weeks after Cycle 1 Day 1 (Cycle length = 28 days)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
percentage of participants
  4-10 weeks after Cycle 6 Day 1 | 22.2 [2.81 to 60.01] | 5.7 [1.18 to 15.66] | 15.7 [7.02 to 28.59] | 31.4 [19.11 to 45.89]
  Year 1 | 33.3 [7.49 to 70.07] | 5.7 [1.18 to 15.66] | 13.7 [5.70 to 26.26] | 21.6 [11.29 to 35.32]
Statistical Analysis 1: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); At 4-10 weeks after Cycle 6 Day 1; Test type: Superiority or Other; Difference in response rates = -15.69, 95% CI 2-sided [-31.87 to 0.49]
Statistical Analysis 2: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); At Year 1; Test type: Superiority or Other; Difference in response rates = -7.84, 95% CI 2-sided [-22.56 to 6.87]

7. Secondary Outcome: Percentage of Participants With Objective Response (OR) According to IRC as Per Lugano Classification, Using PET Scan
Description: OR was defined as CMR or Partial Metabolic Response (PMR). CMR: a score 1 (no uptake above background), 2 (uptake <=mediastinum), or 3 (<mediastinum but <=liver) with or without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites with no new lesions and no evidence of FDG-avid disease in bone marrow. PMR: a score 4 (uptake moderately greater than [>] liver) or 5 (uptake markedly >liver and/or new lesions) with reduced uptake compared with baseline and residual mass(es) of any size on PET 5-PS for lymph nodes and extralymphatic sites with no new lesions and reduced residual uptake in bone marrow compared with baseline. Assessment was performed by an IRC according to Lugano classification using PET scan. 95% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 6-8 weeks after Cycle 6 Day 1 and 48-56 weeks after Cycle 1 Day 1 (Cycle length = 28 days)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
percentage of participants
  6-8 weeks after Cycle 6 Day 1 | 55.6 [21.20 to 86.30] | 21.2 [11.06 to 34.70] | 76.5 [62.51 to 87.21] | 74.5 [60.37 to 85.67]
  Year 1 | 66.7 [29.93 to 92.51] | 32.7 [20.33 to 47.11] | 45.1 [31.13 to 59.66] | 51.0 [36.60 to 65.25]

8. Secondary Outcome: Percentage of Participants With OR According to Investigator as Per Lugano Classification, Using PET Scan
Description: OR was defined as CMR or PMR. CMR: a score 1 (no uptake above background), 2 (uptake <=mediastinum), or 3 (<mediastinum but <=liver) with or without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites with no new lesions and no evidence of FDG-avid disease in bone marrow. PMR: a score 4 (uptake moderately >liver) or 5 (uptake markedly >liver and/or new lesions) with reduced uptake compared with baseline and residual mass(es) of any size on PET 5-PS for lymph nodes and extralymphatic sites with no new lesions and reduced residual uptake in bone marrow compared with baseline. Assessment was performed by Investigator according to Lugano classification using PET scan. 95% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 4-10 weeks after Cycle 6 Day 1 and 48-56 weeks after Cycle 1 Day 1 (Cycle length = 28 days)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
percentage of participants
  4-10 weeks after Cycle 6 Day 1 | 55.6 [21.20 to 86.30] | 28.8 [17.13 to 43.08] | 76.5 [62.51 to 87.21] | 76.5 [62.51 to 87.21]
  Year 1 | 55.6 [21.20 to 86.30] | 21.2 [11.06 to 34.70] | 39.2 [25.84 to 53.89] | 49.0 [34.75 to 63.40]

9. Secondary Outcome: Percentage of Participants With OR According to IRC as Per Lugano Classification, Using CT Scan
Description: OR was defined as CR or Partial Response (PR). CR: reduction of LDi of target nodes/nodal masses to <=1.5 cm, and no extralymphatic sites of disease; absence of non-measured lesions and new lesions; reduction of enlarged organs to normal; and normal/IHC-negative bone marrow morphology. PR: greater than or equal to (>=) 50 percent (%) decrease in sum of the product of the perpendicular diameters (SPD) of up to 6 target measurable nodes and extra-nodal sites; absence/reduction/no increase in size of non-measured lesions; reduction in length of spleen at least >50% beyond normal; and no new lesions. Assessment was performed by an IRC according to Lugano classification using CT scan. 95% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 6-8 weeks after Cycle 6 Day 1 and 48-56 weeks after Cycle 1 Day 1 (Cycle length = 28 days)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
percentage of participants
  6-8 weeks after Cycle 6 Day 1 | 66.7 [29.93 to 92.51] | 30.2 [18.34 to 44.34] | 80.4 [66.88 to 90.18] | 84.3 [71.41 to 92.98]
  Year 1 | 66.7 [29.93 to 92.51] | 22.6 [12.28 to 36.21] | 41.2 [27.58 to 55.83] | 60.8 [46.11 to 74.16]

10. Secondary Outcome: Percentage of Participants With OR According to Investigator as Per Lugano Classification, Using CT Scan
Description: OR was defined as CR or PR. CR: reduction of LDi of target nodes/nodal masses to <=1.5 cm, and no extralymphatic sites of disease; absence of non-measured lesions and new lesions; reduction of enlarged organs to normal; and normal/IHC-negative bone marrow morphology. PR: >=50% decrease in SPD of up to 6 target measurable nodes and extra-nodal sites; absence/reduction/no increase in size of non-measured lesions; reduction in length of spleen at least >50% beyond normal; and no new lesions. Assessment was performed by Investigator according to Lugano classification using CT scan. 95% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 4-10 weeks after Cycle 6 Day 1 and 48-56 weeks after Cycle 1 Day 1 (Cycle length = 28 days)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
percentage of participants
  4-10 weeks after Cycle 6 Day 1 | 55.6 [21.20 to 86.30] | 32.1 [19.92 to 46.32] | 74.5 [60.37 to 85.67] | 78.4 [64.68 to 88.71]
  Year 1 | 55.6 [21.20 to 86.30] | 28.3 [16.79 to 42.35] | 47.1 [32.93 to 61.54] | 49.0 [34.75 to 63.40]

11. Secondary Outcome: Percentage of Participants With OR According to Investigator as Per Lugano Classification, Using PET or CT Scan
Description: OR was defined as CMR/CR or PMR/PR. CMR, CR, PMR, and PR have been defined in previous endpoints, and are not repeated here due to space constraint. Assessment was performed by Investigator according to Lugano classification using PET scan or CT scan (if PET is missing).
Time Frame: Baseline until disease progression or death due to any cause (assessed up to approximately 2.5 years)
Population: ITT population. 'Overall number of participants analyzed'=those evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
percentage of participants | 66.7 [29.93 to 92.51] | 36.5 [23.62 to 51.04] | 80.4 [66.88 to 90.18] | 80.4 [66.88 to 90.18]

12. Secondary Outcome: Duration of Response (DOR) According to Investigator as Per Lugano Classification, Using PET or CT Scan
Description: DOR was defined as time from CMR/CR or PMR/PR until progressive disease (PD) or death due to any cause. CMR, CR, PMR, and PR have been defined in previous endpoints, and are not repeated here due to space constraint. PD: a score 4 (uptake moderately >liver) or 5 (uptake markedly >liver and/or new lesions) with increase in intensity of uptake from baseline on PET 5-PS for individual target nodes/nodal lesions; new FDG-avid foci for extranodal lesions; new FDG-avid foci consistent with lymphoma for new lesions; or new or recurrent FDG-avid foci for bone marrow. Assessment was performed by Investigator according to Lugano classification using PET scan or CT scan (if PET is missing). DOR was calculated using Kaplan-Meier method.
Time Frame: From CMR or PMR until disease progression or death due to any cause (assessed up to approximately 2.5 years)
Population: ITT population. 'Overall number of participants analyzed'=those evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 25 | 47 | 47
months | 32.46 [9.46 to 32.46] | 15.79 [10.15 to 23.49] | 24.87 [12.45 to NA] — Upper limit of 95% CI could not be calculated due to the low number of participants with event. | 15.64 [12.09 to NA] — Upper limit of 95% CI could not be calculated due to the low number of participants with event.
Statistical Analysis 1: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); Stratified Analysis: Strata were disease burden and DOR of prior cancer therapy; Test type: Superiority or Other; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.38 to 1.27] — HR was calculated using Cox regression
Statistical Analysis 2: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); Unstratified Analysis; Test type: Superiority or Other; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.43 to 1.40] — HR was calculated using Cox regression

13. Secondary Outcome: Percentage of Participants With Disease Progression (According to Investigator as Per Lugano Classification, Using PET or CT Scan) or Death
Description: PD: a score 4 (uptake moderately >liver) or 5 (uptake markedly >liver and/or new lesions) with increase in intensity of uptake from baseline on PET 5-PS for individual target nodes/nodal lesions; new FDG-avid foci for extranodal lesions; new FDG-avid foci consistent with lymphoma for new lesions; or new or recurrent FDG-avid foci for bone marrow. Assessment was performed by Investigator according to Lugano classification using PET or CT scan.
Time Frame: Baseline until disease progression or death due to any cause (assessed up to approximately 2.5 years)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
percentage of participants | 44.4 | 86.5 | 41.2 | 52.9

14. Secondary Outcome: Progression-Free Survival (PFS) According to Investigator as Per Lugano Classification, Using PET or CT Scan
Description: PFS was defined as the period from the date of treatment initiation (Safety Run-in and Arm A) or randomization date (Arms B and C) until the date of disease progression, or death due to any cause. PD: a score 4 (uptake moderately >liver) or 5 (uptake markedly >liver and/or new lesions) with increase in intensity of uptake from baseline on PET 5-PS for individual target nodes/nodal lesions; new FDG-avid foci for extranodal lesions; new FDG-avid foci consistent with lymphoma for new lesions; or new or recurrent FDG-avid foci for bone marrow. Assessment was performed by Investigator according to Lugano classification using PET or CT scan. PFS was calculated using Kaplan-Meier method.
Time Frame: Baseline until disease progression or death due to any cause (assessed up to approximately 2.5 years)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
months | 35.09 [12.78 to 35.09] | 6.57 [6.18 to 12.25] | 27.63 [16.07 to NA] — Upper limit of 95% CI could not be calculated due to the low number of participants with event. | 18.43 [16.92 to NA] — Upper limit of 95% CI could not be calculated due to the low number of participants with event.
Statistical Analysis 1: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); Stratified Analysis: Strata were disease burden and PFS of prior cancer therapy; Test type: Superiority or Other; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.38 to 1.24] — HR was calculated using Cox regression
Statistical Analysis 2: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); Unstratified Analysis; Test type: Superiority or Other; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.43 to 1.36] — HR was calculated using Cox regression

15. Secondary Outcome: Percentage of Participants With Disease Progression (According to Investigator as Per Lugano Classification, Using PET or CT Scan), Death, or Start of a New Anti-lymphoma Therapy
Description: as for outcome 13
Time Frame: Baseline until disease progression, death, or start of a new anti-lymphoma therapy whichever occurred first (assessed up to approximately 2.5 years)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
percentage of participants | 44.4 | 86.5 | 41.2 | 52.9

16. Secondary Outcome: Event-Free Survival (EFS) According to Investigator as Per Lugano Classification, Using PET or CT Scan
Description: EFS was defined as the period from the date of treatment initiation (Safety Run-in and Arm A) or randomization date (Arms B and C) to the date of disease progression, death, or start of a new anti-lymphoma therapy whichever occurred first. PD: a score 4 (uptake moderately >liver) or 5 (uptake markedly >liver and/or new lesions) with increase in intensity of uptake from baseline on PET 5-PS for individual target nodes/nodal lesions; new FDG-avid foci for extranodal lesions; new FDG-avid foci consistent with lymphoma for new lesions; or new or recurrent FDG-avid foci for bone marrow. Assessment was performed by Investigator according to Lugano classification using PET or CT scan. EFS was calculated using Kaplan-Meier method.
Time Frame: as for outcome 15
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
months | 35.09 [12.78 to 35.09] | 6.57 [6.18 to 12.25] | 27.63 [16.07 to NA] — Upper limit of 95% CI could not be calculated due to the low number of participants with event. | 18.43 [16.92 to NA] — Upper limit of 95% CI could not be calculated due to the low number of participants with event.
Statistical Analysis 1: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); Stratified Analysis: Strata were disease burden and EFS of prior cancer therapy; Test type: Superiority or Other; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.38 to 1.24] — HR was calculated using Cox regression
Statistical Analysis 2: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); Unstratified Analysis; Test type: Superiority or Other; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.43 to 1.36] — HR was calculated using Cox regression

17. Secondary Outcome: Percentage of Participants Who Died Due to Any Cause
Time Frame: Baseline until death due to any cause (assessed up to approximately 2.5 years
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
percentage of participants | 0 | 5.8 | 2.0 | 3.9

18. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the period from the date of treatment initiation (Safety Run-in and Arm A) or randomization date (Arms B and C) to death due to any cause. For participants who are alive, OS was censored at the last contact. OS was calculated using Kaplan-Meier method.
Time Frame: Baseline until death due to any cause (assessed up to approximately 2.5 years)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Number analyzed (Participants) | 9 | 52 | 51 | 51
months | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to higher number of censored participants. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to higher number of censored participants. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to higher number of censored participants. | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to higher number of censored participants.
Statistical Analysis 1: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); Stratified Analysis: Strata were disease burden and OS of prior cancer therapy; Test type: Superiority or Other; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.04 to 5.37] — HR was calculated using Cox regression
Statistical Analysis 2: Comparison: Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) vs Chemotherapy-Containing Cohort: Arm C (BR); Unstratified Analysis; Test type: Superiority or Other; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.05 to 5.63] — HR was calculated using Cox regression

19. Secondary Outcome: Apparent Clearance (CL) of Venetoclax
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: Pre-dose (within 30 minutes), and 2, 4, 6, 8 hours post-dose on Cycle 1 Day 1; pre-dose (within 30 minutes) on Cycle 1 Days 8, 15, 22; pre-dose (within 30 minutes) and 4 hours post-dose on Day 1 of Cycles 4 and 6 (Cycle length = 28 days)
Population: The data could not be collected as the timepoints for pharmacokinetics collection and the daily dosing of venetoclax did not permit an assessment of CL.
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR)
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Apparent Volume of Distribution (Vd) of Venetoclax
Description: Vd was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: as for outcome 19
Population: The data could not be collected as the timepoints for pharmacokinetics collection and the daily dosing of venetoclax did not permit an assessment of Vd.
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR)
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Venetoclax
Time Frame: as for outcome 19
Population: Pharmacokinetic-evaluable population included all enrolled participants with available pharmacokinetic data for venetoclax.
Measure: Median (Full Range); unit: hours
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR)
Number analyzed (Participants) | 9 | 51 | 46
hours | 8.00 [4.00 to 8.08] | 6.00 [1.95 to 8.18] | 6.21 [1.98 to 9.22]

22. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Venetoclax
Time Frame: as for outcome 19
Population: Pharmacokinetic-evaluable population
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR)
Number analyzed (Participants) | 9 | 51 | 46
nanograms per milliliter (ng/mL) | 1350 (427) | 1220 (478) | 1340 (460)

23. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Last Observed Concentration (AUClast) of Venetoclax
Description: Area under the plasma concentration versus time curve from zero to the last measured concentration (AUClast).
Time Frame: as for outcome 19
Population: Pharmacokinetic-evaluable population
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR)
Number analyzed (Participants) | 9 | 51 | 46
hours*ng/mL | 5310 (1730) | 4950 (1950) | 5500 (2270)

24. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to 8 Hours Post Dose (AUC0-8h) of Venetoclax
Description: Area under the plasma concentration versus time curve from time 0 (pre-dose) to 8 hours post dose (AUC0-8h).
Time Frame: as for outcome 19
Population: Pharmacokinetic-evaluable population. 'Overall number of participants analyzed'=those evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR)
Number analyzed (Participants) | 6 | 30 | 23
hours*ng/mL | 5240 (1860) | 4820 (1980) | 5330 (2270)

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 2.5 years
Description: Safety-evaluable population included participants who received at least one dose of any study treatment.
Arm/Group | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) | Chemotherapy-Containing Cohort: Arm C (BR)
Serious Adverse Events (participants affected / at risk) | 4/9 | 16/52 | 26/49 | 12/50
Other Adverse Events (participants affected / at risk) | 9/9 | 49/52 | 49/49 | 48/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) (N=9) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) (N=52) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) (N=49) | Chemotherapy-Containing Cohort: Arm C (BR) (N=50)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 6 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster disseminated (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 2 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 3 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 3 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Renal stone removal (Surgical and medical procedures) | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 0 | 1 | 0
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 1 | 0 | 0
HERPES SIMPLEX (Infections and infestations) | 0 | 0 | 1 | 0
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy-Containing Cohort:Safety Run-In (Venetoclax + BR) (N=9) | Chemotherapy-Free Cohort: Arm A (Venetoclax + Rituximab) (N=52) | Chemotherapy-Containing Cohort: Arm B (Venetoclax + BR) (N=49) | Chemotherapy-Containing Cohort: Arm C (BR) (N=50)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 19 | 8
Leukopenia (Blood and lymphatic system disorders) | 2 | 5 | 6 | 3
Neutropenia (Blood and lymphatic system disorders) | 5 | 14 | 30 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 7 | 28 | 8
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 2 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 3 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 3 | 0
Vision blurred (Eye disorders) | 1 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 5 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 6 | 6 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 3 | 3
Constipation (Gastrointestinal disorders) | 3 | 5 | 10 | 17
Diarrhoea (Gastrointestinal disorders) | 5 | 21 | 24 | 14
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 3 | 1 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 3 | 2
Nausea (Gastrointestinal disorders) | 7 | 14 | 32 | 23
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 5 | 1
Vomiting (Gastrointestinal disorders) | 4 | 7 | 23 | 13
Asthenia (General disorders) | 1 | 4 | 5 | 4
Catheter site pain (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 5 | 3 | 2
Fatigue (General disorders) | 3 | 13 | 21 | 15
Influenza like illness (General disorders) | 2 | 1 | 2 | 2
Malaise (General disorders) | 0 | 1 | 3 | 0
Mass (General disorders) | 1 | 0 | 0 | 1
Peripheral swelling (General disorders) | 1 | 1 | 2 | 0
Pyrexia (General disorders) | 1 | 5 | 10 | 9
Aspergillus infection (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 6 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 4
Herpes zoster (Infections and infestations) | 1 | 1 | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 3 | 0
Lung infection (Infections and infestations) | 0 | 0 | 4 | 0
Mycobacterium kansasii infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 4 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 4 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 3 | 1
Perineal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 4
Sinusitis (Infections and infestations) | 1 | 3 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 6 | 6 | 4
Urinary tract infection (Infections and infestations) | 1 | 4 | 5 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 18 | 10 | 7
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 5 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 2 | 3
Blood creatinine increased (Investigations) | 0 | 3 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 5
Weight decreased (Investigations) | 1 | 4 | 8 | 0
Weight increased (Investigations) | 0 | 3 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 5 | 10 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 6 | 13 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 6 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 7
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 4 | 8 | 3
Dysgeusia (Nervous system disorders) | 0 | 3 | 3 | 4
Headache (Nervous system disorders) | 3 | 5 | 8 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 2 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 1 | 7 | 2
Dysuria (Renal and urinary disorders) | 2 | 0 | 1 | 2
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 12 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 6 | 2
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 1 | 0 | 2
Hypertension (Vascular disorders) | 1 | 3 | 1 | 2
Hypotension (Vascular disorders) | 2 | 2 | 3 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 4 | 2
COGNITIVE DISORDER (Nervous system disorders) | 1 | 0 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 3
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 0 | 0 | 4 | 2
OEDEMA PERIPHERAL (General disorders) | 0 | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.